CLINICAL TRIAL: NCT01617603
Title: A Comparison Chocolate With and Without High Cocoa Solids in Patients With Type 2 Diabetes in a Randomised Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07.52.NRC
Record Dates: First submitted 2012-06-01; First posted 2012-06-12 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Type 2
Keywords: diabetes type 2; insulin resistance; glycaemic control; Endothelial function; Cocoa Polyphenols
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High polyphenol milk chocolate (Experimental): High polyphenol milk chocolate containing approximately 1 mg/g of epicatechin
  Interventions: Other: Cocoa Polyphenols
- Nestle Noir 70 % chocolate (Active Comparator): Nestle Noir 70 % chocolate containing approximately 1 mg/g of epicatechin
  Interventions: Other: Cocoa Polyphenols
- Low polyphenol milk (Placebo Comparator): Low polyphenol milk control (matched to product 1 as closely as possible for milk content, carbohydrate, fat and calories, made from cocoa butter, sugar, milk powder and small amount of cocoa liquor to improve taste, giving approximately 0.05mg/g epicatechin.
  Interventions: Other: Cocoa Polyphenols

INTERVENTIONS:
Other: Cocoa Polyphenols — 20g/d of product, two active products provide 20 mg/d epicatechin, on visiting occasions, an acute dose of 40g product to be given

SUMMARY:
Type 2 diabetes is being acknowledged as a potential public health time bomb, whose incidence is predicted to double over the next 10 years in the UK, associated with the rise in obesity and increasing sedentary lifestyles. Increased insulin resistance has been shown to be an important feature of type 2 diabetes (especially in those presenting with obesity and in particular visceral or abdominal obesity). Insulin resistance is implicated as a risk factor of cardiovascular disease and may lead to pancreatic dysfunction through increased β-cell stress in the pancreas. A combination of insulin resistance and pancreatic beta cell failure then leads to type 2 diabetes. The main cause of morbidity and mortality in type 2 diabetes is cardiovascular disease as the condition is associated with impaired vascular functioning and increased levels of oxidation markers.

Epidemiological studies suggest dietary flavonoids decrease the risk of death from coronary heart disease, cancer, and stroke. Flavonoid-rich foods include fruits and vegetables as well as tea, red wine, and chocolate. In a cohort of elderly men, cocoa intake was inversely associated with blood pressure and 15-year cardiovascular and all-cause mortality. It has been reported that in healthy humans, consumption of flavanol-rich dark chocolate decreased daytime and night time blood pressure, reduced insulin resistance, and improved nitric oxide dependent vaso-relaxation. Another trial found that cocoa powder increased postprandial insulinaemia in lean young adults. These research papers have led to the hypothesis that chocolate containing high cocoa liquor may help to reduce the risk of developing type 2 diabetes.

This study is design as a double-blind, controlled, single center, randomized, parallel design clinical trial. The primary outcome measure is to compare parameters of insulin resistance and glycaemic control in volunteers with type 2 diabetes after consumption of 3 different chocolates (one dark and two milk chocolates) with a secondary outcome of endothelial function, cholesterol profile and oxidative stress. Subjects will undergo medical screening, anthropometry, physical activity and dietary assessments before randomization.

ELIGIBILITY:
Inclusion criteria:

* The diagnosis of type 2 diabetes will be based on the WHO guidelines. These are 2 fasting plasma glucose readings of greater than 7.0mmoll-1 or 2 random plasma glucose readings >11mmoll-1 in the absence of symptoms or concurrent illness or medication which might lead to hyperglycaemia (e.g. thiazide diuretics). Or one reading meeting the diagnostic level with the presence of symptoms of polyuria, polydipsia, nocturia, fatigue or blurring of vision. The final diagnostic method of diagnosis type 2 diabetes is a positive oral glucose tolerance test (OGTT) using a 75g glucose load. If doubt exists on the diagnosis of diabetes an OGTT will be performed.
* Diabetes managed by diet alone or diet and metformin. If metformin is used the dose should have been stable for a minimum of 3 months prior to the start of the study.
* Hba1c up to and including 9.9%
* Age 45-75
* If female, should be post-menopausal
* BMI 25-39kgm-2
* Patients will have attended a structured group patient education programme (and be on stable medication for hypertension, lipids and gout (if appropriate) for 3 months prior to entry into the study. Subjects will be encouraged to incorporate the chocolate into their diet as advised during the education programme
* Having obtained his/her or his/her legal representative's informed consent.

Exclusion Criteria:

* Patients with concurrent illness or any changes in medication in the last 3 months.
* Patients whose diabetes is managed with TZDs, DPP-IV inhibitors, GLP-1 analogues, insulin or sulphonylureas or prandial regulators
* Patients not wishing to allow disclosure to their GPs.
* Pregnancy
* Hba1c at recruiting stage of >10.0%
* Patient who cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial during the last 3 months prior to the beginning of this study
* Patients who consuming more than 20g/d of chocolate or having a very high polyphenol content of their diet, who are not willing to change their diet
* Patients taking high dose antioxidant supplements including single and multivitamin preparations including A,C,E.
* Women on HRT treatment

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Atkin, MD, Prof, Principal Investigator — Head of Academic Endocrinology, Diabetes & Metabolism; Hull York Medical School; Michael White Diabetes Centre, Hull, UK
Locations (1):
- Endocrinology, Diabetes & Metabolism, Hull York Medical School, Michael White Diabetes Centre, 220-236, Anlaby Road, Hull, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 subjects were recruited. The intention-to-treat (ITT) set comprised of all the subjects who completed V4. One subject joined another trial after recruitment while two other subjects dropped out in course of the trial. These three subjects were not included in the full analysis population. Finally, PP dataset comprised of n = 48.
Pre-assignment Details: Two subjects withdrew their consent quickly after giving it and were replaced so that the total number of recruited subjects was 62. Patients were randomly assigned to one of the three groups using age and gender as the stratification factors. The randomization was performed using the software TRIALSYS (developed internally at Nestlé).
Groups:
- High Polyphenol Milk Chocolate: High polyphenol milk chocolate containing approximately 1 mg/g of epicatechin
  Cocoa Polyphenols : 20g/d of product, two active products provide 20 mg/d epicatechin, on visiting occasions, an acute dose of 40g product to be given
- Low Polyphenol Milk: Low polyphenol milk control (matched to product 1 as closely as possible for milk content, carbohydrate, fat and calories, made from cocoa butter, sugar, milk powder and small amount of cocoa liquor to improve taste, giving approximately 0.05mg/g epicatechin.
  Cocoa Polyphenols : 20g/d of product, two active products provide 20 mg/d epicatechin, on visiting occasions, an acute dose of 40g product to be given
- Nestle Noir 70 % Chocolate: Nestle Noir 70 % chocolate containing approximately 1 mg/g of epicatechin
  Cocoa Polyphenols : 20g/d of product, two active products provide 20 mg/d epicatechin, on visiting occasions, an acute dose of 40g product to be given
Period: Overall Study
Arm/Group | High Polyphenol Milk Chocolate | Low Polyphenol Milk | Nestle Noir 70 % Chocolate
Started | 20 | 21 | 21
Completed | 17 | 19 | 20
Not Completed | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Polyphenol Milk Chocolate | Low Polyphenol Milk | Nestle Noir 70 % Chocolate | Total
Number analyzed (Participants) | 20 | 21 | 21 | 62
Age, Customized [Number; unit: participants]
  <= 45 years | 0 | 0 | 0 | 0
  Between 45 and 75 years | 20 | 21 | 21 | 62
  >=75 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 10 | 31
  Male | 10 | 10 | 11 | 31
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 21 | 21 | 62
HOMA at the begining of product intake [Mean (Inter-Quartile Range); unit: HOMA index] — Baseline HOMA (Homeostatic Model Assessment)index was evaluated at V1 (visit 1) scheduled 28 days after the screening visit (V0) without any chocolate intake. HOMA reflects the resistance to insulin and is obtained from glucose and insulin plasma concentrations at a given sampling timepoint, based on the following formula:
  HOMA = Glucose (in mmol/L) X Insulin ( in mU/L)/ 22.5. Insulin resistance is defined by a HOMA index > 2.4. The highest the HOMA index is, the more pronounced the resistance to insulin is.
  HOMA index | 6.50 [4.14 to 10.21] | 4.63 [2.77 to 7.74] | 4.45 [3.19 to 6.21] | 5.19 [2.77 to 10.21]

OUTCOME MEASURES:

1. Primary Outcome: Difference in Insulin Resistance (HOMA) Between Treatments After 12 Weeks of Product Intake
Description: HbA1c with measurement of plasma glucose and insulin (to determine HOMA index) at the 84th day after product intake minus value at baseline (1st day of product intake. Insulin resistance is defined by a HOMA index > 2.4
Time Frame: 84th day of product intake
Measure: Mean (Inter-Quartile Range); unit: HOMA index
Arm/Group | High Polyphenol Milk Chocolate | Low Polyphenol Milk | Nestle Noir 70 % Chocolate
Number analyzed (Participants) | 17 | 19 | 20
HOMA index | 2.82 [1.93 to 4.14] | 2.21 [1.50 to 3.26] | 2.75 [1.72 to 4.42]

2. Secondary Outcome: Endothelial Function After 12 Weeks of Product Intake
Description: Endothelial function is assessed from arterial stiffness measurements at the 84th day minus the value at baseline (1st day of product intake)
Time Frame: 84th day of product intake
Reporting Status: Not Posted

3. Secondary Outcome: Cholesterol Profile After 12 Weeks of Product Intake
Description: Cholesterol profile is assessed from plasma HDL, LDL and total cholesterol measurements at the 84th day of product intake
Time Frame: 84th day of product intake
Reporting Status: Not Posted

4. Secondary Outcome: Oxidative Stress After 12 Weeks of Product Intake
Description: Oxidative stress is assessed from measurements of plasma markers (High sensitivity CRP, IL-1, IL-6, and alpha-TNF) at the 84th day of product intake
Time Frame: 84th day of product intake
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | High Polyphenol Milk Chocolate | Low Polyphenol Milk | Nestle Noir 70 % Chocolate
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Polyphenol Milk Chocolate (N=20) | Low Polyphenol Milk (N=21) | Nestle Noir 70 % Chocolate (N=21)
Cyst resection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Resection of a papillary cyst in the bladder. Post study SAE, no relationship to the product.
Pacemaker installation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Arrhythmia needing a pacemaker fitting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other